CLINICAL TRIAL: NCT04615585
Title: Evaluation of Local Delivery of Aloe Vera Gel as an Adjunct to Non-surgical Treatment in Patients With Chronic Periodontitis (A Randomized, Clinical Trial)
Brief Title: Evaluation of Local Delivery of Aloe Vera Gel as an Adjunct to Non-surgical Treatment in Patients With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aloevera-chronic periodontitis
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aloe Vera + Scaling and root planing (Experimental)
  Interventions: Other: Aloe vera after SRP
- Scaling and root planing (Active Comparator)
  Interventions: Procedure: Scaling and root planing (SRP)

INTERVENTIONS:
Other: Aloe vera after SRP — Subgingival administration of Aloe vera gel was preceded by flushing the area with saline to wash away any debris. Aloe vera (1cc) gel was applied subgingivally using atraumatic needle. Patients were instructed not to rinse or drink any liquid for at least 30 minutes. The application was performed at baseline and after 1 and 2 weeks.
  Arms: Aloe Vera + Scaling and root planing
Procedure: Scaling and root planing (SRP) — Removal of supragingival and sub-gingival calculus and debris was performed, followed by smoothing root surfaces and removing cementum or dentine that is impregnated with calculus and toxins.
  Arms: Scaling and root planing

SUMMARY:
Aim of the current study was to evaluate the effect of Aloe vera gel as an adjunct to scaling and root planing (SRP) in the management of chronic periodontitis.

DETAILED DESCRIPTION:
The effect of Aloe vera on treatment of chronic periodontitis will be evaluated in a randomized, controlled clinical trial. Thirty patients with mild to moderate chronic periodontitis were divided into 2 groups: group 1 (test): will include 15 patients treated with SRP followed by application of Aloe vera gel in the periodontal pockets at day 1 and after 1 and 2 weeks, and group 2 (control) which includes 15 patients treated with SRP only.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals.
* Patients with mild to moderate chronic periodontitis (CAL 1-4mm) according to the American Academy of Periodontology classification

Exclusion Criteria:

* Smoking and alcoholism.
* Patients with systemic illnesses (i.e., diabetes mellitus, cancer, human immunodeficiency syndrome, bone metabolic diseases, or disorders that compromise wound healing, radiation, or immunosuppressive therapy, conditions leads to xerostomia).
* Patients on any medication affecting the periodontium.
* Lactating, pregnant or menopausal females.
* Patients with parafunctional habits.
* Patients with poor oral hygiene.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Pocket probing depth | up to 9 months
  This was measured using a periodontal probe from the gingival crest to depth of sulcus.
Attachment loss | up to 9 months
  This is measured using a periodontal point. The distance between the cemento-enamel junction and gingival attachment level
Bleeding on probing | up to 9 months
  This is measured using Papillary Bleeding Index (PBI). A periodontal probe is inserted into the gingival sulcus at the base of the papilla on the mesial aspect, and then moved coronally to the papilla tip. This is repeated on the distal aspect of the papilla. The intensity of any bleeding is recorded as:
  Score 0 - no bleeding; Score 1 - A single discreet bleeding point; Score 2 - Several isolated bleeding points or a single line of blood appears; Score 3 - The interdental triangle fills with blood shortly after probing; Score 4 - Profuse bleeding occurs after probing; blood flows immediately into the marginal sulcus.
Plaque index | up to 9 months
  This will be assessed on 4 surfaces of 6 index teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four in order to give the plaque index for the tooth with the following scores and criteria. 0:No plaque, 1: A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface. 2: Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye. 3: Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Gingival index | up to 9 months
  This will be assessed on 4 surfaces of 6 index teeth. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3. The scores from the four areas of the tooth are added and divided by four in order to give the gingival index for the tooth with the following scores and criteria. 0= Normal gingiva; 1= Mild inflammation - slight change in color and slight edema but no bleeding on probing; 2= Moderate inflammation - redness, edema and glazing, bleeding on probing; 3= Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma E Tayeb, BDS, Principal Investigator — Faculty of Dentistry, Alexandria University, Egypt; Mohy E El Rashidy, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Rania A Fahmy, PhD, Study Director — Faculty of Dentistry, Alexandria University, Egypt; Mohamed S Abdel Gaffar, PhD, Study Director — Faculty of Pharmacy, Alexandria University, Egypt; Reham A Abo Elwafa, PhD, Study Director — Faculty of Medicine, Alexandria University, Egypt
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Background] Wiebe CB, Putnins EE. The periodontal disease classification system of the American Academy of Periodontology--an update. J Can Dent Assoc. 2000 Dec;66(11):594-7. PMID 11253351
- [Background] Salgado AD, Maia JL, Pereira SL, de Lemos TL, Mota OM. Antiplaque and antigingivitis effects of a gel containing Punica granatum Linn extract: a double-blind clinical study in humans. J Appl Oral Sci. 2006 Jun;14(3):162-6. doi: 10.1590/s1678-77572006000300003. PMID 19089066
- [Background] Botelho MA, Nogueira NA, Bastos GM, Fonseca SG, Lemos TL, Matos FJ, Montenegro D, Heukelbach J, Rao VS, Brito GA. Antimicrobial activity of the essential oil from Lippia sidoides, carvacrol and thymol against oral pathogens. Braz J Med Biol Res. 2007 Mar;40(3):349-56. doi: 10.1590/s0100-879x2007000300010. PMID 17334532
- [Background] Davis RH, Leitner MG, Russo JM, Byrne ME. Wound healing. Oral and topical activity of Aloe vera. J Am Podiatr Med Assoc. 1989 Nov;79(11):559-62. doi: 10.7547/87507315-79-11-559. PMID 2607423
- [Background] Ahmadi A. Potential prevention: Aloe vera mouthwash may reduce radiation-induced oral mucositis in head and neck cancer patients. Chin J Integr Med. 2012 Aug;18(8):635-40. doi: 10.1007/s11655-012-1183-y. Epub 2012 Aug 2. PMID 22855041
- [Background] Singh N, Hebbale M, Mhapuskar A, Ul Nisa S, Thopte S, Singh S. Effectiveness of Aloe Vera and Antioxidant along with Physiotherapy in the Management of Oral Submucous Fibrosis. J Contemp Dent Pract. 2016 Jan 1;17(1):78-84. doi: 10.5005/jp-journals-10024-1806. PMID 27084867
- [Background] Babaee N, Zabihi E, Mohseni S, Moghadamnia AA. Evaluation of the therapeutic effects of Aloe vera gel on minor recurrent aphthous stomatitis. Dent Res J (Isfahan). 2012 Jul;9(4):381-5. PMID 23162576
- [Background] Bhalang K, Thunyakitpisal P, Rungsirisatean N. Acemannan, a polysaccharide extracted from Aloe vera, is effective in the treatment of oral aphthous ulceration. J Altern Complement Med. 2013 May;19(5):429-34. doi: 10.1089/acm.2012.0164. Epub 2012 Dec 16. PMID 23240939